CLINICAL TRIAL: NCT03312738
Title: A Randomized, Double-blind, Placebo Controlled, Phase II Study of Everolimus in Combination With Exemestane in the Treatment of Chinese Postmenopausal Women With Estrogen Receptor Positive, HER-2 Negative, Locally Advanced, Recurrent, or Metastatic Breast Cancer After Recurrence or Progression on Prior Letrozole or Anastrozole
Brief Title: A Study of Everolimus Plus Exemestane in Chinese Postmenopausal Women With Estrogen Receptor Positive, Locally Advanced, Recurrent, or Metastatic Breast Cancer After Recurrence or Progression on Non-steroidal Aromatase Inhibitor
Acronym: BOLERO-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001Y2202
Record Dates: First submitted 2017-09-15; First posted 2017-10-18 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-04

CONDITIONS: Advanced Breast Cancer
Keywords: everolimus; exemestane; advanced Breast Cancer; non-steroidal aromatase inhibitors; breast carcinoma; breast cancer; breast lump; HER2 negative; breast cancer progression
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Everolimus + Exemestane (Experimental): Participants received everolimus as a continuous oral daily dose of 10 mg and exemestane as a continuous oral daily dose of 25 mg
  Interventions: Drug: Everolimus; Drug: Exemestane
- Placebo + Exemestane (Active Comparator): Participants received placebo as a continuous oral daily dose and exemestane as a continuous oral daily dose of 25 mg
  Interventions: Drug: Exemestane; Drug: Everolimus Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus was formulated as tablets of 5 mg strength and was packaged into blister packs . Everolimus (two 5 mg tablets daily) was administered in a blinded manner by continuous oral daily dosing.
  Other Names: RAD001
  Arms: Everolimus + Exemestane
Drug: Exemestane — Commercially available exemestane was supplied as 25 mg tablets. Exemestane was administered as continuous oral daily dose of 25 mg tablets.
Drug: Everolimus Placebo — Placebo was formulated to be indistinguishable from the everolimus tablets. Matching placebo (two tablets daily) was administered in a blinded manner by continuous oral daily dosing.
  Arms: Placebo + Exemestane

SUMMARY:
This study aimed at evaluating the safety and efficacy of everolimus plus exemestane in Chinese postmenopausal women with ER+ HER2- locally advanced, recurrent, or metastatic breast cancer after recurrence or progression on letrozole or anastrozole.

DETAILED DESCRIPTION:
This was a multicenter, double-blind, randomized, placebo-controlled, phase II study evaluating treatment with everolimus (10 mg daily) in combination with exemestane (25 mg daily) vs placebo in combination with exemestane (25 mg daily) in Chinese postmenopausal women with locally advanced, recurrent or metastatic ER+ HER2- breast cancer refractory to non-steroidal aromatase inhibitors.

Randomized participants started the study treatment at Cycle 1 Day 1, and were treated continuously until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death or discontinuation from treatment for any other reason.

After end of treatment, all participants were followed up for safety up to 30 days after last dose of study treatment (exemestane and/or everolimus/placebo). All participants were followed for survival status at least every 3 months after treatment discontinuation unless they discontinued due to death, consent withdrawal or lost to follow-up

If a participants permanently discontinued study treatment for reasons other than disease progression, death, lost to follow-up, or withdrawal of consent to efficacy follow-up then they entered the post-treatment efficacy follow-up period until disease progression, death, lost to follow-up or withdrawal of consent for efficacy follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Chinese Postmenopausal women with ER+ HER2- locally advanced, recurrent, or metastatic breast cancer. Locally advanced breast cancer must not be amenable to curative treatment by surgery or radiotherapy.
* Histological or cytological confirmation of estrogen-receptor positive (ER+) breast cancer
* Postmenopausal women. Postmenopausal status was defined either by:

  * Prior bilateral oophorectomy
  * Or age ≥60
  * Or age < 60 and amenorrhea for 12 or more months
* Recurrence or progression on prior NSAI was defined as:

  * Recurrence while on, or within one year (12 months) of end of adjuvant treatment with letrozole or anastrozole
  * Or Progression while on or within one month (30 days) of the end of prior treatment with letrozole or anastrozole
* Radiological or objective evidence of recurrence or progression on or after the last systemic therapy prior to enrollment
* Patient had as per RECIST 1.1

  * measurable disease or non-measurable lytic or mixed (lytic + blastic) bone lesions in the absence of measurable disease.
  * non-measurable lytic or mixed (lytic + blastic) bone lesions in the absence of measurable disease.
* Patient was able to swallow and retain oral medication
* Patient met the hematologic and biochemistery laboratory values at the screening visit
* Patient had a WHO performance status ≤2
* Written informed consent obtained prior to any screening procedures

Exclusion Criteria:

* HER2-overexpressing patients by local laboratory testing (IHC 3+ staining or in situ hybridization positive), based on the most recent test.
* Patients who had received more than one chemotherapy line for ABC
* Patients with symptomatic visceral disease and candidates to chemotherapy
* Patients with only non-measurable lesions other than lytic or mixed (lytic and blastic) bone metastasis (e.g. pleural effusion, ascites etc.)
* Patients receiving concomitant immunosuppressive agents or chronic corticosteroids used at the time of study entry except topical applications, inhaled sprays, eye drops or local injections.
* Uncontrolled diabetes mellitus as defined by HbA1c >7% despite adequate therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- China (14):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Shao ZM, Cai L, Wang S, Hu X, Shen K, Wang H, Li H, Feng J, Liu Q, Cheng J, Wu X, Wang X, Li H, Luo T, Liu J, Amin K, Slimane K, Qiao Y, Liu Y, Tong Z. BOLERO-5: a phase II study of everolimus and exemestane combination in Chinese post-menopausal women with ER + /HER2- advanced breast cancer. Discov Oncol. 2024 Jun 21;15(1):237. doi: 10.1007/s12672-024-01027-8. PMID 38904918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 15 investigative sites in China
Pre-assignment Details: The screening period began once patients had signed the study informed consent. All screening/baseline evaluations were performed within maximum 21 days prior to the first dose of study treatment
Period: Overall Study
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Started | 80 | 79
Completed | 0 | 0
Not Completed | 80 | 79
Not completed — Progressive disease | 58 | 67
Not completed — Patient/guardian decision | 13 | 5
Not completed — Adverse Event | 5 | 3
Not completed — Protocol deviation | 2 | 0
Not completed — Technical problems | 0 | 1
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane | Total
Number analyzed (Participants) | 80 | 79 | 159
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (9.14) | 56.3 (8.43) | 56.4 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 79 | 159
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 80 | 79 | 159

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Based on Local Radiology Review of Tumor Assessment
Description: PFS was defined as time from the date of randomization to the date of first documented progression or death due to any cause. A patient who had not progressed or died at the date of the analysis cut-off or received another anticancer therapy had their PFS censored at the time of the last adequate tumor evaluation before the earlier of the cut-off date or the anticancer therapy date. Disease progression was assessed using the local investigator's tumor assessment per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
  The distribution of PFS was estimated using the Kaplan-Meier method. Cox regression model stratified by randomization stratification factors was used to estimate the hazard ratio (HR) of PFS, along with 90% CI. As this was an estimation based approach, no p-value was provided.
Time Frame: From randomization up to date of first documented progression or death, assessed up to approximately 3.5 years
Population: Full Analysis Set (FAS) including all subjects to whom study treatment was assigned by randomization.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Months | 7.4 [5.5 to 9.2] | 2.0 [1.9 to 3.6]
Statistical Analysis 1: Comparison: Everolimus + Exemestane vs Placebo + Exemestane; Test type: Other; Hazard Ratio (HR) = 0.53, 90% CI 2-sided [0.40 to 0.71]

2. Secondary Outcome: Progression-free Survival (PFS) Based on Blinded Independent Review Committee (BIRC) Assessment
Description: PFS was defined as time from the date of randomization to the date of first documented progression or death due to any cause. A patient who had not progressed or died at the date of the analysis cut-off or received another anticancer therapy had their PFS censored at the time of the last adequate tumor evaluation before the earlier of the cut-off date or the anticancer therapy date. Disease progression was assessed using the BIRC tumor assessment per RECIST 1.1.
  The distribution of PFS was estimated using the Kaplan-Meier method. Cox regression model stratified by randomization stratification factors was used to estimate the hazard ratio (HR) of PFS, along with 90% CI. As this was an estimation based approach, no p-value was provided.
Time Frame: From randomization up to date of first documented progression or death, assessed up to approximately 1.8 years
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Months | 7.4 [5.5 to 9.3] | 3.1 [1.9 to 3.7]
Statistical Analysis 1: Comparison: Everolimus + Exemestane vs Placebo + Exemestane; Test type: Other; Hazard Ratio (HR) = 0.46, 90% CI 2-sided [0.32 to 0.67]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to date of death due to any cause. If the participant was alive at the date of the analysis cut-off or lost to follow-up, then OS was censored at the last contact date prior to data cutoff date.
  The distribution of OS was estimated using the Kaplan-Meier method. Cox regression model stratified by randomization stratification factors was used to estimate the hazard ratio (HR) of OS, along with 90% CI. As this was an estimation based approach, no p-value was provided.
Time Frame: From randomization to date of death, up to approximately 3.8 years
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Months | 26.1 [20.2 to 33.7] | 22.7 [18.6 to 37.8]
Statistical Analysis 1: Comparison: Everolimus + Exemestane vs Placebo + Exemestane; Test type: Other; Hazard Ratio (HR) = 1.14, 90% CI 2-sided [0.69 to 1.89]

4. Secondary Outcome: Overall Response Rate (ORR) Based on Local Radiology Review of Tumor Assessment
Description: ORR was defined as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR) according to RECIST using local radiologist's/investigator's tumor assessment. ORR was estimated and the exact binomial 90% CI was reported by treatment arm.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 3.5 years
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Percentage of participants | 10.0 [5.1 to 17.3] | 2.5 [0.5 to 7.8]

5. Secondary Outcome: Overall Response Rate (ORR) Based on BIRC Assessment
Description: ORR was defined as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR) according to RECIST using BIRC assessment. ORR was estimated and the exact binomial 90% CI was reported by treatment arm.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 1.8 years
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Percentage of participants | 8.8 [4.2 to 15.8] | 2.5 [0.5 to 7.8]

6. Secondary Outcome: Clinical Benefit Rate (CBR) Based on Local Radiology Review of Tumor Assessment
Description: CBR was defined as the percentage of patients with best overall response of CR, PR or an overall lesion response of stable disease (SD) or Non-CR/Non-progressive disease with duration of 24 weeks or longer according to RECIST 1.1 using local radiologist's/investigator's tumor assessment. CBR was estimated and the exact binomial 90% CI was reported by treatment arm.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 3.5 years
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Percentage of participants | 42.5 [33.1 to 52.3] | 16.5 [10.0 to 24.9]

7. Secondary Outcome: Clinical Benefit Rate (CBR) Based on BIRC Assessment
Description: CBR was defined as the percentage of patients with best overall response of CR, PR or an overall lesion response of stable disease (SD) or Non-CR/Non-progressive disease with duration of 24 weeks or longer according to RECIST 1.1 using BIRC assessment. CBR was estimated and the exact binomial 90% CI was reported by treatment arm.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease.
Time Frame: Up to approximately 1.8 years
Population: FAS including all subjects to whom study treatment was assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Percentage of participants | 31.3 [22.7 to 40.8] | 11.4 [6.1 to 19.0]

8. Secondary Outcome: Time to Response (TTR) Based on Local Radiology Review of Tumor Assessment
Description: TTR was defined as the time between date of randomization until first documented response (CR or PR) according to RECIST 1.1 using local radiologist's/investigator's tumor assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 3.5 years
Population: Participants in the FAS with a confirmed CR or PR as per local radiologist's/investigator's tumor assessment.
Measure: Median (Full Range); unit: Days
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 8 | 2
Days | 84.5 [51 to 162] | 53.0 [52 to 54]

9. Secondary Outcome: Time to Response (TTR) Based on BIRC Assessment
Description: TTR was defined as the time between date of randomization until first documented response (CR or PR) according to RECIST 1.1 using BIRC assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 1.8 years
Population: Participants in the FAS with a confirmed CR or PR as per BIRC assessment
Measure: Median (Full Range); unit: Days
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 7 | 2
Days | 57.0 [15 to 224] | 81.5 [52 to 111]

10. Secondary Outcome: Duration of Response (DOR) Based on Local Radiology Review of Tumor Assessment
Description: DOR was defined as the time from date of first documented CR or PR to date of first documented disease progression or death due to any cause, according to RECIST 1.1 using local radiologist's/investigator's tumor assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first documented response to date of first documented disease progression or death, assessed up to approximately 3.5 years
Population: Participants in the FAS with a confirmed CR or PR as per local radiologist's/investigator's tumor assessment
Measure: Median (Full Range); unit: Days
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 8 | 2
Days | 243.5 [110 to 624] | 561.5 [282 to 841]

11. Secondary Outcome: Duration of Response (DOR) Based on BIRC Assessment
Description: DOR was defined as the time from date of first documented CR or PR to date of first documented disease progression or death due to any cause, according to RECIST 1.1 using BIRC assessment.
  CR: Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm.
  PR: At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From date of first documented response to date of first documented disease progression or death, assessed up to approximately 1.8 years
Population: Participants in the FAS with a confirmed CR or PR as per BIRC assessment
Measure: Median (Full Range); unit: Days
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 7 | 2
Days | 148.0 [57 to 281] | 279.0 [221 to 337]

12. Secondary Outcome: Time to Definitive Deterioration of the Eastern Cooperative Oncology Group Performance Status (ECOG PS) by at Least One Category of the Score From Baseline
Description: ECOG PS is a measure of functional status with scores ranging from 0 (fully active) to 5 (dead). Deterioration was considered definitive if no improvements in the ECOG PS status were observed after an instance of deterioration. Death was considered as worsening of the ECOG PS if it occurred close to the last assessment, where "close" is defined as twice the planned period between two assessments. Participants who died after more than twice the planned period between two assessments were censored at the date of their last assessment before the cut-off. Participants receiving any further anticancer therapy prior to definitive worsening were censored at their date of last assessment prior to start of therapy. Participants that had not worsened were censored at the date of last assessment prior to cut off. Time to definitive deterioration was estimated using the Kaplan-Meier method.
Time Frame: From randomization up to definitive deterioration of the ECOG PS by one categotu of the score, assessed up to approximately 3.5 years
Population: FAS including all subjects to whom study treatment was assigned by randomization
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Months | NA [NA to NA] — Not estimable (NA) due to the low number of participants with deterioration of ECOG PS | NA [NA to NA] — Not estimable (NA) due to the low number of participants with deterioration of ECOG PS

13. Secondary Outcome: Everolimus Predose Concentration (Cmin)
Description: Blood samples were collected to assess everolimus predose concentration (Cmin) at steady state at Cycle 1 Week 4 (any day during week 4). Steady-state was defined as having no dose adjustment/interruption of everolimus and exemestane in the previous 4 days prior to the day of the pre-dose PK sample collection.
  Everolimus concentrations were determined in the whole blood by a liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. The method has a lower limit of quantitation (LLOQ) of 0.3 ng/mL for everolimus. Values below the LLOQ were set to 0.
Time Frame: Predose on Cycle 1 Week 4 ( each cycle is defined as 4 weeks)
Population: All subjects with an evaluable everolimus concentration at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/mililiter (ng/mL)
Arm/Group | Everolimus + Exemestane
Number analyzed (Participants) | 70
nanogram/mililiter (ng/mL) | 16.5 (59.1)

14. Secondary Outcome: Everolimus Concentration at 2 Hours Post Dose (C2h)
Description: Blood samples were collected to assess everolimus concentration at 2 hours post dose (C2h) at steady state at Cycle 1 Week 4 (any day during week 4) Steady-state was defined as having no dose adjustment/interruption of everolimus and exemestane in the previous 4 days prior to the day of the pre-dose PK sample collection.
  Everolimus concentrations were determined in the whole blood by a liquid chromatography with tandem mass spectrometry (LC-MS/MS) method. The method has a LLOQ of 0.3 ng/mL for everolimus. Values below the LLOQ were set to 0.
Time Frame: Two hours post everolimus administration on Cycle 1 Week 4 ( each cycle is defined as 4 weeks)
Population: All subjects with an evaluable everolimus concentration at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Everolimus + Exemestane
Number analyzed (Participants) | 71
ng/mL | 44.2 (57.8)

15. Secondary Outcome: Exemestane Predose Concentration (Cmin)
Description: Blood samples were collected to assess exemestane predose concentration (Cmin) at steady state at Cycle 1 Week 4 (any day during week 4). Steady-state was defined as having no dose adjustment/interruption of everolimus and exemestane in the previous 4 days prior to the day of the pre-dose PK sample collection.
  Exemestane concentrations were determined in the whole blood by a liquid chromatography with LC-MS/MS method. The method has a LLOQ of 20 pg/mL for exemestane. Values below the LLOQ were set to 0.
Time Frame: Predose of exemestane on Cycle 1 Week 4 ( each cycle is defined as 4 weeks)
Population: All subjects with an evaluable exemestane concentration at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/mililiter (pg/mL)
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 71 | 71
picogram/mililiter (pg/mL) | 737 (74.2) | 502 (48.7)

16. Secondary Outcome: Exemestane Concentration at 2 Hours Post Dose (C2h)
Description: Blood samples were collected to assess exemestane concentration at 2 hours post dose (C2h) at steady state at Cycle 1 Week 4 (any day during week 4) Steady-state was defined as having no dose adjustment/interruption of everolimus and exemestane in the previous 4 days prior to the day of the pre-dose PK sample collection.
  Exemestane concentrations were determined in the whole blood by a liquid chromatography with LC-MS/MS method. The method has a LLOQ of 20 pg/mL for exemestane. Values below the LLOQ were set to 0.
Time Frame: Two hours post exemestane administration on Cycle 1 Week 4 ( each cycle is defined as 4 weeks)
Population: All subjects with an evaluable exemestane concentration at the specified time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 72 | 73
pg/mL | 20500 (97.1) | 14300 (71.6)

17. Secondary Outcome: Estradiol Levels After 4 Weeks of Study Treatment
Description: Blood samples were collected to assess estradiol levels after 4 weeks of study treatment. Estradiol was determined in plasma using competitive immunoassay. The method has a LLOQ of 1.952 pg/mL for estradiol. Values below the LLOQ were set to 0.
Time Frame: Baseline, and at Cycle 1 Week 4 prior to any study drug (each cycle is defined as 4 weeks)
Population: All subjects with evaluable estradiol concentrations at the specified time points
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 72 | 70
pg/mL
  Baseline | 5.98 (10.5) | 5.38 (10.4)
  Week 4 | 3.98 (7.77) | 3.77 (6.80)

18. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study medication to 30 days after the last dose of study medication for a maximum duration of approximately 3.5 years Post-treatment survival follow-up deaths were collected after 30 days post-treatment, for a maximum duration of approximately 3.8 years All deaths refer to the sum of on-treatment and post-treatment deaths
Time Frame: On-treatment deaths: Up to 3.5 years. Post-treatment survival follow-up deaths: Up to 3.8 years
Population: Safety set including all subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Exemestane | Placebo + Exemestane
Number analyzed (Participants) | 80 | 79
Participants
  On-treatment deaths | 3 | 2
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 73 | 75
  Post-treatment survival follow-up deaths | 41 | 43
  All deaths | 44 | 45

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment to 30 days after last dose of study medication (on-treatment), up to approx. 3.5 years. Deaths were collected in the post treatment survival follow up from 31 days after last dose of study medication until the end of the study, up to approx. 3.8 years. These are not considered AEs
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
Groups:
- Everolimus + Exemestane (On-treatment): AEs collected during on-treatment period (up to 30 days post-treatment)
- Placebo + Exemestane (On-treatment): AEs collected during on-treatment period (up to 30 days post- treatment)
- Everolimus + Exemestane (Post-treatment Survival Follow-up); Placebo + Exemestane (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 31 post- treatment). No AEs were collected during this period
Arm/Group | Everolimus + Exemestane (On-treatment) | Placebo + Exemestane (On-treatment) | Everolimus + Exemestane (Post-treatment Survival Follow-up) | Placebo + Exemestane (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 3/80 | 2/79 | 41/73 | 43/75
Serious Adverse Events (participants affected / at risk) | 18/80 | 10/79 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 79/80 | 62/79 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane (On-treatment) (N=80) | Placebo + Exemestane (On-treatment) (N=79) | Everolimus + Exemestane (Post-treatment Survival Follow-up) (N=0) | Placebo + Exemestane (Post-treatment Survival Follow-up) (N=0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | NA | NA
Cardiac failure (Cardiac disorders) | 1 | 0 | NA | NA
Vomiting (Gastrointestinal disorders) | 1 | 0 | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | NA | NA
Pyrexia (General disorders) | 1 | 0 | NA | NA
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | NA | NA
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | NA | NA
Herpes virus infection (Infections and infestations) | 1 | 0 | NA | NA
Pneumonia (Infections and infestations) | 6 | 0 | NA | NA
Subcutaneous abscess (Infections and infestations) | 1 | 0 | NA | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Neutrophil count decreased (Investigations) | 1 | 0 | NA | NA
Diabetic ketosis (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Renal failure (Renal and urinary disorders) | 1 | 0 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Exemestane (On-treatment) (N=80) | Placebo + Exemestane (On-treatment) (N=79) | Everolimus + Exemestane (Post-treatment Survival Follow-up) (N=0) | Placebo + Exemestane (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 26 | 10 | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 10 | 3 | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 5 | 0 | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0 | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0 | NA | NA
Aphthous ulcer (Gastrointestinal disorders) | 12 | 2 | NA | NA
Diarrhoea (Gastrointestinal disorders) | 10 | 3 | NA | NA
Mouth ulceration (Gastrointestinal disorders) | 19 | 3 | NA | NA
Nausea (Gastrointestinal disorders) | 10 | 6 | NA | NA
Stomatitis (Gastrointestinal disorders) | 28 | 5 | NA | NA
Toothache (Gastrointestinal disorders) | 6 | 1 | NA | NA
Vomiting (Gastrointestinal disorders) | 10 | 4 | NA | NA
Asthenia (General disorders) | 5 | 3 | NA | NA
Chest discomfort (General disorders) | 2 | 4 | NA | NA
Malaise (General disorders) | 9 | 0 | NA | NA
Oedema peripheral (General disorders) | 10 | 0 | NA | NA
Pyrexia (General disorders) | 6 | 3 | NA | NA
Pneumonia (Infections and infestations) | 11 | 3 | NA | NA
Upper respiratory tract infection (Infections and infestations) | 8 | 6 | NA | NA
Urinary tract infection (Infections and infestations) | 8 | 0 | NA | NA
Alanine aminotransferase increased (Investigations) | 28 | 14 | NA | NA
Aspartate aminotransferase increased (Investigations) | 38 | 15 | NA | NA
Bilirubin conjugated increased (Investigations) | 0 | 4 | NA | NA
Blood albumin decreased (Investigations) | 5 | 0 | NA | NA
Blood alkaline phosphatase increased (Investigations) | 5 | 4 | NA | NA
Blood bilirubin increased (Investigations) | 3 | 5 | NA | NA
Blood cholesterol increased (Investigations) | 10 | 2 | NA | NA
Blood creatine phosphokinase increased (Investigations) | 13 | 3 | NA | NA
Blood creatinine increased (Investigations) | 6 | 4 | NA | NA
Blood glucose increased (Investigations) | 5 | 1 | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 8 | 3 | NA | NA
Blood triglycerides increased (Investigations) | 5 | 0 | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 14 | 6 | NA | NA
Low density lipoprotein increased (Investigations) | 9 | 1 | NA | NA
Neutrophil count decreased (Investigations) | 13 | 8 | NA | NA
Platelet count decreased (Investigations) | 14 | 5 | NA | NA
Weight decreased (Investigations) | 23 | 3 | NA | NA
Weight increased (Investigations) | 1 | 4 | NA | NA
White blood cell count decreased (Investigations) | 16 | 5 | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 17 | 4 | NA | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 21 | 0 | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 36 | 6 | NA | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 3 | NA | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 | 3 | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 5 | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 1 | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2 | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 0 | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5 | NA | NA
Headache (Nervous system disorders) | 2 | 5 | NA | NA
Insomnia (Psychiatric disorders) | 8 | 2 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 6 | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 14 | 0 | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | NA | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5 | 1 | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3 | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 11 | 1 | NA | NA
Hypertension (Vascular disorders) | 6 | 2 | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03312738/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03312738/SAP_001.pdf